CLINICAL TRIAL: NCT01968876
Title: Is a Smartphone Application Effective as an Oral Medication Adherence Aid
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study had a minor contingency that could not be resolved with the IRB.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202266
Record Dates: First submitted 2013-10-10; First posted 2013-10-24 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Hypertension; Diabetes; Dyslipidemia
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): The control group will not use the medication adherence app
- Medication Adherence Smartphone App (Experimental): The experimental group will receive the medication adherence app on their smartphone and will have their entire outpatient medication list pushed to the application. Text message reminders will be sent to their phones at the appropriate times.
  Interventions: Other: Medication Adherence Smartphone App

INTERVENTIONS:
Other: Medication Adherence Smartphone App — MyMedSchedule is a consumer-grade smartphone application currently available on various marketplaces of the Android and iOS platforms that acts as a portal to the free service MyMedSchedule.com website. It can interface with the MedActionPlan discharge planning tool for providers by automatically populating fields, allowing medication lists to be pushed to a subject's MyMedSchedule account, allowing the input of complex medication regimens, and aiding in medication reconciliation. A MyMedSchedule account can be setup with the patient's name, date of birth, allergies, emergency contact, healthcare providers, insurance plan information, and complete medication list. Medication dose and refill reminders can be set and sent through short message service (SMS) text message or e-mail. SMS text message reminders will be used for this study.
  Other Names: MyMedSchedule
  Arms: Medication Adherence Smartphone App

SUMMARY:
This research will act as a pilot study that will be conducted to determine the effectiveness of a smartphone medication adherence application on adherence to oral hypertensive, diabetic, and dyslipidemic medications using a prospective randomized design. Subjects will be recruited from the University of Arkansas for Medical Sciences (UAMS) Internal Medicine Clinic North, and the study data will be collected using only subject self-reports and subject pharmacy records.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age
* Provide informed consent
* Prescribed an oral medication indicated for hypertension, diabetes, or dyslipidemia during 12 weeks pre-enrollment
* Own a smartphone (Android or iOS) with unlimited text messaging, email access, and app store access
* Oral confirmation that the subject has not previously used a medication adherence app
* Able to consult with a pharmacy or medical student during the recruitment process for purposes of consent, data collection, and/or medication reconciliation, and/or MyMedSchedule registration

Exclusion Criteria:

* Severely impaired vision
* Reside in a nursing home
* Non-ambulatory/bedridden
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of pills taken over number of pills prescribed at 4 weeks | Change from baseline to 4 weeks
Change from baseline in number of pills taken over number of pills prescribed at 12 weeks | Change from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul H Anderson, Principal Investigator — University of Arkansas
Locations (3):
- United States (3):
  - Internal Medicine Clinic North; University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Remedy Drug, Little Rock, Arkansas
  - Internal Medicine Clinic West; University of Arkansas for Medical Sciences, Little Rock, Arkansas